CLINICAL TRIAL: NCT06788223
Title: Intraoperative Identification of Parathyroid Adenomas Using PTeye™ and FLUOBEAM® LX: a Prospective Cohort Study
Acronym: PTeye
Status: Active, not recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Papavramidis Theodossis, Professor, Aristotle University Of Thessaloniki
Other Study IDs: PTeye
Record Dates: First submitted 2025-01-02; First posted 2025-01-23 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Primary Hyperparathyroidism Due to Adenoma
MeSH Terms: conditions — Parathyroid Neoplasms | interventions — Parathyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PTeye: Localizing Parathyroid adenoma with the PTeye device during parathyroidectomy
  Interventions: Device: Parathyroidectomy
- Fluobeam: Localizing Parathyroid adenoma with the Fluobeam/ Fluoptics device
  Interventions: Device: Parathyroidectomy

INTERVENTIONS:
Device: Parathyroidectomy — Parathyroidectomy under general anesthesia

SUMMARY:
The goal of this observational study is to evaluate the efficacy of PTeyeTM device to confirm a parathyroid adenoma on a visually suspected tissue in comparison with the FLUOBEAM®LX device. The main questions it aims to answer is:

Is the PTeyeTM device effective in identifying the presence of a parathyroid adenoma? Which autofluorecence device (PTeye or FLUOBEAM®LX) is more effective in confirming the presence of a parathyroid adenoma? Participants will undergo parathyroidectomy under general anesthesia. During the procedure visually suspected tissue for parathyroid adenoma will be evaluated with the PTeye or FLUOBEAM®LX device for the presence of an adenoma (minute 0). Tissue will be reevaluated on minutes 1, 3, and 5 and before excision.

DETAILED DESCRIPTION:
Objective: PTeye™ and FLUOBEAM® LX use autofluorescence to confirm visually suspected parathyroid tissue. Real-time intraoperative identification of parathyroid glands can be achieved by the application of both devices. The aim of the present study is to evaluate and compare the efficacy of PTeye™ and FLUOBEAM® LX in identifying parathyroid adenomas.

Methods: Patients undergoing parathyroidectomy due to a parathyroid adenoma will be enrolled prospectively in this study and will be randomly included to Group A (PTeye™) or Group B (FLUOBEAM® LX). After intraoperative identification of parathyroid adenomas and before tissue dissection (minute 0), the efficacy of both devices to confirm the adenomas will be evaluated. Re-evaluation will take place in minutes 1, 3 and 5 during tissue dissection and before adenoma excision.

ELIGIBILITY:
Inclusion Criteria:

- Patients with Primary parathyroidism with parathyroid adenoma

Exclusion Criteria:

* Parathyroid Hyperplasia,
* Secondary hyperparathyroidism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary hyperparathyroidism and parathyroid adenoma, fulfilling the AAES guidelines indications for parathyroidectomy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Identification of the parathyroid adenoma | The minute of the identification of the parathyroid adenoma (minute 0). Reevaluation in minutes 1, 3, and 5 during tissue dissection and before excision.
  The percentage of adenomas identified by each device is assessed after intraoperative identification of parathyroid adenomas and before tissue dissection (minute 0).
  The same percentage will be re-evaluated on minutes 1, 3 and 5 during tissue dissection and before adenoma excision.

CONTACTS AND LOCATIONS:
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code